CLINICAL TRIAL: NCT03842540
Title: The Share Health Study: Teens Social Connections and Health (Phase 2)
Brief Title: The Share Health Study: Teen Social Connections and Health (Phase 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #16-19206 App v1.15
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Contraception
Keywords: LARC; Contraceptive decision-making; Diffusion of Innovations

STUDY DESIGN:
Intervention Model Description: SpeakOut: Empowering Teen to Teen Social Communication About Highly Effective Contraception (Also Known As: The Share Health Study: Teen Social Connections and Health) (Phase 2)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SpeakOut Intervention (Experimental): Primary participants will be randomized to this arm or the Alcohol Control Arm at the time of enrollment. Secondary participants will be assigned to this arm if the primary participant whom initially told them about the study is in this arm. Primary participants in this arm will receive the SpeakOut intervention and will complete surveys on their contraceptive knowledge, attitudes, behaviors, and social communication at baseline, three months, and nine months. Secondary participants in this arm will complete similar surveys at baseline, three months, and nine months.
  Note: Secondary participants will not receive intervention, but will be assessed on outcomes that may have been affected as a result of social communication with primary participants.
  Interventions: Behavioral: SpeakOut
- PartyWise Intervention (Active Comparator): Primary participants will be randomized to this arm or the SpeakOut Intervention Arm at the time of enrollment. Secondary participants will be assigned to this arm if the primary participant whom initially told them about the study is in this arm. Primary participants in this arm will receive the Alcohol Control Intervention on the day of enrollment, and will complete surveys on their contraceptive knowledge, attitudes, behaviors, and social communication at baseline, three months, and nine months. Secondary participants in this arm will complete similar surveys at baseline, three months, and nine months.
  Note: Secondary participants will receive an intervention, but will be assessed on outcomes that may have been affected as a result of social communication with primary participants.
  Interventions: Behavioral: PartyWise

INTERVENTIONS:
Behavioral: SpeakOut — SpeakOut aims to increase social communication about contraception between adolescent IUD and implant users and their peers. SpeakOut has four components:
  1. Coaching session. Research staff will deliver a script to encourage recipients to share information about their contraceptive method with peers.
  2. Digital materials for recipients to keep and/or share with friends.
  3. Websites with information and resources. Staff will refer recipients to a website, either SpeakOutIUD.org or SpeakOutImplant.org, which contain information about their method.
  4. Text messages with information about recipients' method and about how to share their experience. Recipients will be given the opportunity to sign up for text messages that will be sent for 8 weeks following receipt of SpeakOut.
  Arms: SpeakOut Intervention
Behavioral: PartyWise — The active comparator intervention is an alcohol assessment and education intervention using an SBIRT (Screening, Brief Intervention, and Referral to Treatment) framework. Staff will ask two screening questions developed by the National Institute on Alcohol Abuse and Alcoholism (NIAAA) and the American Academy of Pediatrics to screen for adolescents potentially at risk. Using a script based on tenets of motivational interviewing to assess alcohol related consequences, the staff will guide teens in identifying personally relevant motivators for healthier behaviors, assess readiness to change, and offer educational materials and referrals.
  Arms: PartyWise Intervention

SUMMARY:
The purpose of this study is to determine whether delivery of SpeakOut, a behavioral intervention to increase social communication about long-acting reversible contraceptive (LARC) methods among adolescents, is associated with increased contraceptive use among the social contacts of SpeakOut recipients.

The investigators will conduct a cluster randomized controlled trial of SpeakOut with adolescent LARC users and their female peers. Over three years, SpeakOut will be implemented in eight partner clinics. IUD and implant users aged 15 to 19 will be recruited online and invited to enroll in the evaluation study as "primary" participants and receive either SpeakOut or a control intervention about alcohol use called PartyWise. The social contacts of primary participants will be asked to enroll in the study as "secondary" participants. The study's primary outcome will be the proportion of sexually-active secondary participants who are using any contraceptive method at 9-month follow-up.

DETAILED DESCRIPTION:
Teen pregnancy results from under-use contraception by sexually active teens. Social networks are important influences on teen contraceptive knowledge and use. Encouraging social communication to increase knowledge and acceptability of LARC among female adolescents can increase use of contraception.

The Share Health Study is a cluster randomized control trial, randomized at the primary participant level. Primary participants will be randomized to receive either SpeakOut or a control intervention about alcohol use (PartyWise) immediately before intervention delivery. A cluster consists of primary participants and the secondary participants recruited to the study via a specialized snowball sampling procedure carried out with the assistance of the primary participant, described below.

Primary participant procedures

Adolescents ages 15-19 years old who are using an IUD or implant will be recruited through targeted social media advertisements.

After providing consent, each primary participant will complete a baseline survey collecting demographic information and asking about contraceptive knowledge, attitudes, use, and social communication as well as drug and alcohol behaviors.

Primary participants will be randomized to receive either SpeakOut or the control intervention and receive the assigned intervention immediately after randomization by phone. Each delivery session lasts about 10 minutes, and both SpeakOut and control sessions will be audio-recorded and observed for quality and fidelity measurement by UC Davis staff. Primary participants will be instructed to ask up to five social contacts if they would be willing to participate in the study and will send them a link to an online screener and survey.

The SpeakOut intervention is informed by the Theory of Diffusion of Innovation and aims to increase social communication about IUDs and implants between adolescent IUD and implant users and their peers. The intervention is comprised of four components:

1. A one-on-one communication coaching session for teen IUD and implant users. Contracted staff will deliver an educational script by phone to review effective communication strategies and encourage primary participants to share information about their contraceptive method of choice with peers, to the extent they feel comfortable.
2. Method-specific digital materials for recipients to keep and/or share with friends. Staff will provide pamphlets designed to a) deliver evidence-based information about their method, and b) facilitate communication about their choice with social contacts, including about their experience with the method and their reasons for choosing it.
3. Method-specific websites with information and resources. Staff will refer teens to a website, either SpeakOutIUD.org or SpeakOutImplant.org, which contain information about their method, including the information contained in the pamphlets, resources related to sharing their experience with their peers, and links to online information provided by the National Campaign through their online birth control support network, Bedsider.org. This includes location and contact information for clinics that provide LARC, videos featuring individuals who use these methods, and the opportunity to explore multiple methods using Bedsider's method comparison feature.
4. Method-specific text messages with information about recipients' method and about how to share their experience. Recipients will be given the opportunity to sign up for text messages that will be sent every week for 8 weeks following receipt of SpeakOut in clinic. These texts will provide evidence-based information about use of the method (e.g., address concerns about menstrual spotting), in order to promote accurate knowledge and facilitate ongoing use of the method, and provide reinforcement of the value of sharing their story.

The counterfactual intervention for SpeakOut - called PartyWise - is an alcohol assessment and education intervention using an SBIRT (Screening, Brief Intervention, and Referral to Treatment) framework. SBIRT is an evidence-based practice model aimed at preventing problematic use and identifying potential abuse and dependency issues. The approach includes an early intervention focus so that individuals with non-dependent alcohol use are identified and supported in moving towards avoidance or reduction in alcohol use and educated about ways to minimize harm. The participant will be asked two screening questions electronically, developed by the National Institute on Alcohol Abuse and Alcoholism (NIAAA) and the American Academy of Pediatrics to screen for adolescents potentially at risk. Using a script based on tenets of motivational interviewing to assess alcohol related consequences, the study staff will guide teens in identifying personally relevant motivators for healthier behaviors, assess readiness to change, and offer educational materials. Participants who receive this intervention will have the option to sign up for text messages with additional information about alcohol consumption for 8 weeks following enrollment. Motivational Interviewing is patient-centered and utilizes the adolescent's own intrinsic motivations for change. It is based on the stages of change theoretical model in which readiness to make changes resides on a continuum and the client and counselor together explore how to help the client make the changes she is ready for or address how to help the client move towards increased readiness to make positive changes. With the participant's permission, delivery of this intervention will be audio-recorded by contracted staff.

For both experimental and control interventions, staff will offer participants the opportunity to receive text message content via email, if they have an email address and no mobile phone that receives text messages.

3 months after enrollment, contracted staff and/or research staff will contact primary participants by phone call, text, and/or e-mail and ask them to complete the first follow-up survey over the phone or online. The survey will include questions about contraceptive knowledge, attitudes, and use as well as drug and alcohol behaviors.

9 months after enrollment, contracted staff or research staff will contact primary participants by phone, text, and/or e-mail and ask them to complete the second follow-up survey over the phone or by-email. The survey will include questions about contraceptive knowledge, attitudes, and use as well as drug and alcohol behaviors.

Secondary participant procedures

Potential secondary participants will be approached by the primary participant. Primary participants will ask for potential secondary participants' to participate in the study by sending them a link to a website with study information, a screening tool to assess the secondary participants' eligibility, and a baseline survey for eligible participants.

Eligible participants will link to an electronic consent with more information about the study. If they are interested, they will indicate their consent by selecting a check box on an electronic consent form in Qualtrics, a secure survey program with electronic consent capability, on their device.

If the secondary participant consents electronically, they will be linked to the baseline survey collecting demographic information and asking about contraceptive knowledge, attitudes, use, and social communication, as well as drug and alcohol behaviors.

Three months after enrollment of their primary participant, contracted staff or research staff will contact secondary participants by phone, text, and/or e-mail and ask them to complete the first follow-up survey electronically or by phone. The survey will include questions about contraceptive knowledge, attitudes, use, and social communication as well as drug and alcohol behaviors. Contracted staff or research staff will attempt to reach primary participants for up to one month following the 3-month post-enrollment date.

Nine months after enrollment of their primary participant, contracted staff or research staff will contact secondary participants by phone call, text, and/or e-mail and ask them to complete the second follow-up survey over the phone or by-email. The survey will include questions about contraceptive knowledge, attitudes, and use as well as drug and alcohol behaviors.

ELIGIBILITY:
Inclusion Criteria:

Primary participants:

* Age 15 to 19
* Female
* Able to speak and read English or Spanish easily
* Uses an IUD or implant for birth control
* Is comfortable with close friend knowing that they use an IUD or implant
* Can think of at least one friend or family member they would be comfortable asking to join a study about health topics like birth control and alcohol use
* If minor, lives in state where they are able to consent for reproductive health services

Secondary participants:

* 15 to 20 years old
* Female
* Able to speak and read English or Spanish easily
* Was listed as a social contact by a primary participant at enrollment, and can name that primary participant at screening
* If minor, lives in state where they are able to consent for reproductive health services.

Exclusion Criteria:

Primary participants:

* Previous enrollment as a primary or secondary participant in the study
* Pregnant at baseline

Secondary participants:

* Pregnant at baseline
* Previous enrollment as a primary secondary participant in the study*

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1099 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Contraceptive use among secondary participants | Up to 9 months
  Proportion of secondary participants reporting use of any contraceptive method in follow-up surveys.
  Outcome is dichotomous (Yes, USING contraception/No, NOT using contraception) and based on responses to PI-authored Survey item 1: What birth control method (s) are you currently using to prevent pregnancy? (Check all that apply of the following 11 response options)
  "Yes, USING contraception" defined as those who check any of the following:
  1. Pill (Birth control pill)
  2. Patch (Birth control patch)
  3. Ring ("Nuvaring")
  4. Shot ("Depo")
  5. Hormonal IUD (Mirena, Liletta, or Skyla)
  6. Non-hormonal IUD (Paragard or "copper T")
  7. Implant (Nexplanon or Implanon, rod under skin of arm)
  8. Condoms
     "No, NOT using contraception" defined as those who do not check items 1-8 above, whether or not they check any of the following response options:
  9. Withdrawal/pulling out
  10. Other
  11. I am not currently using a method to prevent pregnancy

SECONDARY OUTCOMES:
Implant initiation (among all secondary participants, those recently sexually active, and ever sexually active) | Up to 9 months
  Proportion of secondary participants reporting initiation of implant in follow-up surveys.
  Outcome is dichotomous (Yes, initiated implant/No, did not initiate implant) and based on responses to PI-authored Survey item 1: What birth control method (s) are you currently using to prevent pregnancy? (Check all that apply of the following 11 response options)
  "Yes, initiated IUD" defined as those who check the following:
  7. Implant (Nexplanon or Implanon, rod under skin of arm)
  "No, not did not initiate IUD" defined as those who do not check item 7, whether or not they check any other responses.
IUD initiation (ie current IUD use among those not using an IUD at baseline) among secondary participants | Up to 9 months
  Proportion of secondary participants reporting initiation of IUD in follow-up surveys.
  Outcome is dichotomous (Yes, initiated IUD/No, did not initiate IUD) and based on responses to PI-authored Survey item 1: What birth control method (s) are you currently using to prevent pregnancy? (Check all that apply of the following 11 response options)
  "Yes, initiated IUD" defined as those who check the following:
  5.Hormonal IUD (Mirena, Liletta, or Skyla) 6.Non-hormonal IUD (Paragard or "copper T")
  "No, not did not initiate IUD" defined as those who do not check items 5 or 6, whether or not they check any other responses.
Initiation of contraceptive used by primary participant among secondary participants reporting sexual active | Up to 9 months
  Proportion of secondary participants reporting initiation of the LARC method used by their cluster primary participant in follow-up surveys.
  Outcome is dichotomous (Yes, initiated primary's LARC/No, did not initiate primary's LARC) and based on responses to PI-authored Survey item 1: What birth control method (s) are you currently using to prevent pregnancy? (Check all that apply of the following 11 response options)
  "Yes, initiated primary's LARC" defined as those who check the following (IUD or implant, depending on what method primary used at baseline):
  5.Hormonal IUD (Mirena, Liletta, or Skyla) 6.Non-hormonal IUD (Paragard or "copper T") 7. Implant (Nexplanon or Implanon, rod under skin of arm)
  "No, not did not initiate primary's LARC" defined as those who do not check item 5, 6, or 7 (depending on primary's method), whether or not they check any other responses.
Positive attitudes towards cluster primary participant's LARC method among secondary participants | Up to 9 months
  Mean score of secondary participants on PI-authored scale measure; "Overall, how would you rate each of the following as a birth control method for yourself, even if you've never used it? Please choose a number from 0 to 10 based on your opinion of each method, using the following scale. If you haven't heard of a method, choose "Never heard of it."
  * IUD
  * Implant (Nexplanon or Implanon, rod under skin of arm)
  Scale presented, range 0 - 10 (or never heard of it)
  0= Terrible method 10= Great method
Knowledge of cluster primary participant's LARC use among secondary participants | Up to 9 months
  Proportion of secondary participants giving correct response on to PI-authored item about primary participant's LARC use.
  Dichotomous; "What birth control method do you think [user] is using?" Yes=correct answer (IUD or implant) No=Incorrect answer Combined with info on primary participant's method use from primary participant follow-up survey.
Knowledge of LARC methods among secondary participants | Up to 9 months
  Mean score of secondary participants on knowledge inventory derived from National Survey of Reproductive and Contraceptive Knowledge. Score 0-6 combining correct True/False responses to six items about either IUD or implant, depending on cluster primary participant's method. Higher score represents higher knowledge.
Positive social communication about LARC method between primary and secondary participants | Up to 9 months
  Proportion of secondary respondents giving response of 4 or 5 on PI-authored 5-point Likert scale of agreement/disagreement with statement of positive content of discussion.
  Dichotomized; "Think about when you have talked with [user] about the [hormonal IUD/non-hormonal IUD/implant]. How much do you agree or disagree with the following statements about talking to [user] about the [IUD/implant]?
  [User] told me good things about the [IUD/implant]."
  (Response options 01. Strongly disagree / 02. Disagree / 03. Neither agree nor disagree / 04. Agree / 05. Strongly agree)
  Yes=response 4 or 5 No=any other responses
Negative social communication about LARC method between primary and secondary participants | Up to 9 months
  Proportion of secondary respondents giving response of 4 or 5 on 5-point Likert scale of agreement/disagreement with statement of positive content of discussion.
  Dichotomized; "Think about when you have talked with [user] about the [hormonal IUD/non-hormonal IUD/implant]. How much do you agree or disagree with the following statements about talking to [user] about the [IUD/implant]?
  [User] told me bad things about the [IUD/implant]."
  (Response options 01. Strongly disagree / 02. Disagree / 03. Neither agree nor disagree / 04. Agree / 05. Strongly agree)
  Yes=response 4 or 5 No=any other responses
Condom use at last sexual intercourse among sexually active secondary participants | Up to 9 months
  Proportion of sexually secondary participants reporting condom use at last intercourse in response to PI-authored survey item:
  Dichotomized (Yes, used condoms/No, did not use condoms); "The last time you had vaginal sex, did you use any of these methods of birth control?
  Check all that apply:
  1. Pill (Birth control pill)
  2. Patch (Birth control patch)
  3. Ring ("Nuvaring")
  4. Shot ("Depo")
  5. Hormonal IUD (Mirena, Liletta, or Skyla)
  6. Non-hormonal IUD (Paragard or "copper T")
  7. Implant (Nexplanon or Implanon, rod under skin of arm)
  8. Condoms
  9. Withdrawal 10. Other
  Yes=response 8 checked No=response 8 not checked
Diagnosis of sexually transmitted infection among secondary participants | Up to 9 months
  Proportion of secondary participants reporting diagnosis of STI and STI type in PI-authored items:
  Has a doctor or nurse told you [in the past 3 months/in the past 6 months] that you had a sexually transmitted infection? 1, Yes 0, No 2, Don't know
  What infections have you had [in the past 3 months/in the past 6 months]?
  1. Chlamydia
  2. Gonorrhea
  3. Trichomoniasis (or Trich)
  4. Other a. What infection(s) have you had in the past [3/6] months?
Initiation of sexual activity among secondary participants | Up to 9 months
  Proportion of secondary participants reporting ever having had sexual intercourse in response to PI-authored item in follow-up surveys.
  Dichotomous; "Have you ever had vaginal sex? (By vaginal sex we mean, penis in vagina)" Yes=1 No=0 Don't know=2, will be dropped
Pregnancy among secondary participants | Up to 9 months
  Proportion of secondary participants reporting pregnancy during study period in response to PI-authored item in follow-up surveys.
  Dichotomous (Yes/No); "Have you ever been pregnant (even if you did not give birth)?" (If yes) "How many times have you been pregnant?
IUD continuation among primary participants | Up to 9 months
  Proportion of primary participants reporting continuation of their IUD in follow-up surveys.
  Outcome is dichotomous (Yes, continuing IUD/No, not continuing IUD) and based on responses to PI-authored Survey item 1: What birth control method (s) are you currently using to prevent pregnancy? (Check all that apply of the following 11 response options)
  "Yes, continuing IUD" defined as those who check the following:
  5.Hormonal IUD (Mirena, Liletta, or Skyla) 6.Non-hormonal IUD (Paragard or "copper T")
  "No, not continuing IUD" defined as those who do not check items 5 or 6, whether or not they check any other responses.
Implant continuation among primary participants | Up to 9 months
  Proportion of primary participants reporting continuation of their implant in follow-up surveys.
  Outcome is dichotomous (Yes, continuing implant/No, not continuing implant) and based on responses to PI-authored Survey item 1: What birth control method (s) are you currently using to prevent pregnancy? (Check all that apply of the following 11 response options)
  "Yes, continuing implant" defined as those who check the following:
  7.Implant (Nexplanon or Implanon, rod under skin of arm)
  "No, not continuing implant" defined as those who do not check item 7, whether or not they check any other responses.
Positive attitudes towards LARC method among primary participants | Up to 9 months
  Mean score of secondary participants on PI-authored scale measure; "Overall, how would you rate each of the following as a birth control method for yourself, even if you've never used it? Please choose a number from 0 to 10 based on your opinion of each method, using the following scale. If you haven't heard of a method, choose "Never heard of it."
  * IUD
  * Implant (Nexplanon or Implanon, rod under skin of arm)
  Scale presented, range 0 - 10 (or never heard of it)
  0= Terrible method 10= Great method
Knowledge of LARC method among primary participants | Up to 9 months
  Mean score of primary participants on knowledge inventory derived from National Survey of Reproductive and Contraceptive Knowledge. Score 0-6 combining correct True/False responses to six items about either IUD or implant, depending on participant's method. Higher score represents higher knowledge.
Initiation of social communication about LARC method among primary participants | Up to 9 months
  Proportion of secondary participants giving positive response to PI-authored item in in follow-up surveys.
  Dichotomous (Yes/No); "Have you talked about birth control with a female friend or family member in the past month?"
Pregnancy among primary participants | Up to 9 months
  Proportion of primary participants reporting pregnancy during study period in response to PI-authored item in follow-up surveys.
  Dichotomous (Yes/No); "Have you ever been pregnant (even if you did not give birth)?" (If yes) "How many times have you been pregnant?
Risk of unintended pregnancy (ie sex without contraception) | Up to 9 months
  Proportion of primary and secondary participants reporting risky sex during study period in response to Office of Adolescent Health- authored item.
  Dichotomous (Yes/No): "In the past three/six months, have you had vaginal sex without using at least one of these methods of birth control?
  * Pill (Birth control pill)
  * Patch (Birth control patch)
  * Ring ("Nuvaring")
  * Shot ("Depo")
  * IUD (Hormonal IUD Mirena, Liletta, or Skyla OR Non-hormonal IUD Paragard or "copper T")
  * Implant (Nexplanon or Implanon, rod under skin of arm)
  * Condoms"
Alcohol use | Up to 9 months
  Mean days of alcohol use as reported in response to item derived from Youth Risk Behavior Survey.
Knowledge of binge-drinking behaviors | Up to 9 months
  Proportion of participants giving correct responses to knowledge items of what constitutes binge drinking, including sex differences in binge drinking. Items derived from the Youth Risk Behavior Survey.
Acceptability of SpeakOut | Up to 9 months
  Proportion of participants giving positive responses to PI-authored items to understand participants' experience with and opinion of different intervention components of SpeakOut. Will be examined among both primary and secondary participants.
Acceptability of PartyWise [control intervention] | Up to 9 months
  Proportion of participants giving positive responses to PI-authored items to understand participants' experience with and opinion of different intervention components of PartyWise. Will be examined among both primary and secondary participants.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Dehlendorf, MD, MAS, Principal Investigator — University of California, San Francisco; Kathleen Tebb, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Kathleen Tebb, San Francisco, California, United States

REFERENCES:
- [Derived] Schwarz EB, Chatterton B, Fix M, Tebb K, Rodriguez F, Tancredi DJ, Muriki M, Satterfield J. Remotely Educating Young Women About Alcohol: A Randomized Trial of the PartyWise Intervention. J Womens Health (Larchmt). 2022 Aug;31(8):1179-1187. doi: 10.1089/jwh.2021.0285. Epub 2022 Feb 28. PMID 35230177